CLINICAL TRIAL: NCT01678235
Title: The Impact Of Insulin Glulisine In Comparison With Aspart On Postprandial Glycemia After The High-Glycemic Index Meal In Children With Type 1 Diabetes - Cross-Over Double-Blind, Randomized Clinical Trial.
Brief Title: Insulin Glulisine and Aspart in Postprandial Glycemic Control After High-GI Meal in Children With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Glulisine_Aspart
Record Dates: First submitted 2012-08-28; First posted 2012-09-03 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2012-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes; insulin pump; glulisine; aspart; glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — insulin glulisine; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLU_ASP (Experimental): Pre-breakfast insulin was given as a standard bolus 15 minutes before the high-glycemic index meal (cornflakes and milk). The carbo-insulin ratio on both study days was identical to the patient's ratio when entering trial.
  First day: insulin glulisine
  Second day: insulin aspart
  Interventions: Drug: Insulin glulisine; Drug: Insulin aspart
- ASP_GLU (Experimental): Pre-breakfast insulin was given as a standard bolus 15 minutes before the high-glycemic index meal (cornflakes and milk). The carbo-insulin ratio on both study days was identical to the patient's ratio when entering trial.
  First day: insulin aspart
  Second day: insulin glulisine
  Interventions: Drug: Insulin glulisine; Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin glulisine
  Other Names: Apidra®
Drug: Insulin aspart
  Other Names: NovoRapid®

SUMMARY:
The aim of this study is to determine whether insulin glulisine is more effective in postprandial glycemic control than insulin aspart after the H-GI meal in children with type 1 diabetes (T1DM) treated with insulin pump (CSII).

DETAILED DESCRIPTION:
Some studies have suggested that insulin glulisine (GLU) has a slightly faster onset of action compared with insulin aspart (ASP). Meals of high glycemic index (H-GI) have distinct effect on postprandial glycaemia (PPG).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* CSII for at least 3 months
* Duration of diabetes > 1 years
* Informed consent

Exclusion Criteria:

* Concomitant dietary restrictions (e.g. celiac disease or food allergy)
* Diabetes related complications
* Baseline hyperglycemia >150 mg/dl
* Any disease judged by the investigator to affect the trial

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemia | baseline, 30, 60, 90, 120 and 180 minutes after the breakfast

SECONDARY OUTCOMES:
Hypoglycemia episodes | 3-h study period
  Hypoglycemia was defined as a PG concentration below 65 mg/dl with or without symptoms
Glucose Area Under the Curve (AUC) | 3-h study period
  based on continuous glucose monitoring system
Mean amplitude of glycemic excursion (MAGE) | 3-h study period
Difference between the maximum and baseline glycemia | 3-h study period

OTHER OUTCOMES:
Questionnaire: Glycemic Index Knowledge | each subject was asked to fullfill the questionnaire before entering the study (day one)

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Dżygało, MD, Principal Investigator — Department of Pediatrics, Medical University of Warsaw, Poland
Locations (1):
- Department of Pediatrics, Medical University of Warsaw, Poland, Warsaw, Poland

REFERENCES:
- [Result] Dzygalo K, Szypowska A. Impact of insulins glulisine and aspart on postprandial glycemia after a high-glycemic index meal in children with type 1 diabetes. Eur J Endocrinol. 2014 Mar 8;170(4):539-45. doi: 10.1530/EJE-13-0696. Print 2014 Apr. PMID 24412929